CLINICAL TRIAL: NCT03195764
Title: A Phase I Safety and Tolerability Study of T-1101 (Tosylate) as a Oral Powder for Constitution (OPC) in Patients With Advanced Refractory Solid Tumors
Brief Title: Safety and Tolerability Study for T-1101 (Tosylate) to Treat Advanced Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated before the primary endpoint (determination of MTD) was reached because the OPC form is to be replaced with the newly developed capsule form in all subsequent clinical trials.
Sponsor: Taivex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAI-001
Record Dates: First submitted 2017-05-08; First posted 2017-06-22 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Advanced Refractory Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-1101 (Tosylate) (Experimental)
  Interventions: Drug: T-1101 (Tosylate)

INTERVENTIONS:
Drug: T-1101 (Tosylate) — T-1101 (Tosylate) powder in bottle

SUMMARY:
T-1101 (Tosylate) is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by Taivex Therapeutics Corp. T-1101 (Tosylate) is a potent anti-cancer agent in numerous human cancer cell lines. In addition, oral administration of T-1101 (Tosylate) showed tumor growth inhibition in different mouse xenograft models of human cancers. In this study, safety, tolerability and PK of T-1101 (Tosylate) will be evaluated and also the recommended dose and regimen(s) to initiate Phase 2 will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor eligibility:

   * Histologically confirmed advanced malignancies refractory to standard active treatment.
   * Solid tumors that have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy.
2. Able, in the investigator's opinion, to have a life expectancy of more than 3 months.
3. Female or male, 20 years of age or older.
4. ECOG performance status 0 or 1.
5. Resolution of all acute toxic effects of prior therapy or surgical procedures to no more than grade 1 (except alopecia).
6. Adequate organ function as defined by the following criteria:

   * Serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN), or ALT ≤ 5 x ULN if liver tumor is present.
   * Total serum bilirubin ≤1.5 x ULN
   * WBC ≥ 4000/µL with an absolute neutrophil count (ANC) ≥1500/µL
   * Platelets ≥ 100,000/µL
   * Hemoglobin ≥ 9.0 g/dL
   * CCr ≥ 50 mL/min
7. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Major surgery (as defined by investigator) within 4 weeks of starting treatment.
2. Extensive radiation therapy or systemic cytotoxic chemotherapy within 4 weeks before starting study treatment or target therapy within 2 weeks of starting study treatment.
3. Current treatment on clinical trial or within 4 weeks of completion of clinical trial for another investigation drug.
4. Documented or suspicious brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.
5. Any of the following occurs within 6 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
6. Ongoing cardiac dysrhythmias of NCI CTCAE grade 2, or atrial fibrillation of any grade.
7. Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
8. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
9. Known human immunodeficiency virus infection.
10. Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to the use of highly effective contraception during the period of therapy. Highly effective method of birth control is defined as one that results in a low failure rate (i.e. less than 1 percent per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, or a vasectomized partner. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the patient inappropriate for entry into this study.
12. Patients with active infection should be excluded.
13. Positive test for hepatitis B (HBsAg) or hepatitis C (anti-HCV antibody).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of T-1101 (Tosylate) in Participants with Advanced Cancers Refractory to Standard Therapy | The first 21-day cycle
  MTD is highest dose level in which 6 patients have been treated with at most 1 experiencing dose limiting toxicity (DLT).
  When following toxicity events occur within the first 21-day cycle, these toxicity will be defined as DLT.
  1. Hematological toxicities : prolonged grade 4 neutropenia for >7 days, grade 3 febrile neutropenia (an ANC < 1000/mm3 with a single temperature of > 38.3°C or a sustained temperature of > 38°C for more than 1 hour), grade 4 febrile neutropenia (febrile neutropenia with life-threatening consequences; urgent intervention indicated), grade 3 neutropenia with grade 3 infection and grade 3 thrombocytopenia with bleeding or grade 4 lasting 7 days.
  2. Non-hematological toxicities: grade 3 or 4 toxicities, Nausea and vomiting or diarrhea must persist at grade 3 or 4 despite maximal medical therapy.
  The above toxicities will be graded according to the NCI CTCAE v4.03.

SECONDARY OUTCOMES:
Pharmacokinetics: Peak maximum plasma concentration (Cmax) and minimum plasma concentration (Cmin) of T-1101 (Tosylate) and its metabolites | Selected time points during first 21-day cycle
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) to the time of the last measurable concentration and to infinity of T-1101 (Tosylate) and its metabolites | Selected time points during first 21-day cycle
  Area under the plasma concentration versus time curve to the time of the last measurable concentration (AUC0-last) of T-1101 (Tosylate) and its metabolites will be estimated using non-compartmental analysis. If data permit, area under the plasma concentration versus time curve to infinity (AUC0-∞) will be also estimated.
Pharmacokinetics: Time to maximum plasma concentration (Tmax) and terminal half-life (T½) of T-1101 (Tosylate) and its metabolites | Selected time points during first 21-day cycle
  Time to maximum plasma concentration (Tmax) of T-1101 (Tosylate) and its metabolites will be estimated using non-compartmental analysis. If data permit, terminal elimination half-life (T½ ) will be also estimated.
Pharmacokinetics: Oral plasma clearance (CL/F) of T-1101 (Tosylate) and its metabolites | Selected time points during first 21-day cycle
Pharmacokinetics: Apparent volume of distribution (Vd/F) of T-1101 (Tosylate) and its metabolites | Selected time points during first 21-day cycle
Clinical Tumor Response of T-1101 (Tosylate) in Participants with Advanced Cancers | Up to 2 years
  Categorization of response based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No